CLINICAL TRIAL: NCT03241901
Title: "Aiming at Prolonging the Therapeutic Life Span of Artemisinin-based Combination Therapies (ACT) in an Era of Imminent Plasmodium Falciparum Resistance in Bagamoyo District, Tanzania - New Strategies With Old Tools"
Brief Title: "Prolonging the Therapeutic Life Span of Artemisinin-based Combination Therapies (ACT) in Bagamoyo District, Tanzania"
Acronym: ALU-PQ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: Uppsala University (Other); Karolinska Institutet (Other); The University of Western Australia (Other)
Responsible Party: Principal Investigator, Dr. Lwidiko Edward, Medical Doctor, Muhimbili University of Health and Allied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No. 01.05.2017
Record Dates: First submitted 2017-07-05; First posted 2017-08-08 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Malaria,Falciparum
Keywords: Artemether-Lumefantrine, Primaquine
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination; Primaquine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Due to the objectives of the study, the identity of test and control treatments will be known only to investigators, research staff, but NOT patients. The following study procedures will be in place to ensure single-blind administration of study treatments.
  1. Access to the randomization code will be strictly controlled.
  2. A taste-matching agent for the placebo.
  3. Packaging and labeling of test and control treatments will be identical to maintain the blind.
  During the study, the blind may be broken only in emergencies when knowledge of the patient's treatment group is necessary for further patient management. When possible, the Investigator should discuss the emergency with the Medical Monitor prior to un-blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 Days Artemether-Lumefantrine + Placebo (Active Comparator): Oral tablets of artemether-lumefantrine (20-120mg):
  1. tablet for 5-14kg;
  2. tablets for 15-24 kg;
  3. tables for 25 - 34kg and
  4. tablets for above 35 Kg. The full course of treatment is 6-doses for 3 days given twice daily, at 0, 8, 24, 36, 48, 60 with the dose being given as directly observed therapy.
  Oral placebo after completion of the standard 3 days-six dose regimen. A fatty snack (biscuits) will be administered together with all artemether-lumefantrine doses to optimize absorption.
  Interventions: Drug: Artemether-Lumefantrine Tab 20-120mg; Other: Placebo
- 6Days Artemether/Lumefantrine+Primaquine (Experimental): Artemether-lumefantrine (20-120mg) twice daily for 6 days according to body weight as in the active comparator arm.
  And in addition to that, , a single 0.25 mg/kg primaquine dose (Primaquine phosphate) will be administered concomitantly with the last (i.e. twelfth) artemether-lumefantrine dose. Primaquine will be prepared and administered in an aqueous solution.
  Interventions: Drug: Artemether-Lumefantrine Tab 20-120mg; Drug: Primaquine Phosphate 0.25 mg/kg

INTERVENTIONS:
Drug: Artemether-Lumefantrine Tab 20-120mg — Artemether-Lumefantrine Tablet 20-120mg
  Other Names: ALU
Drug: Primaquine Phosphate 0.25 mg/kg — Primaquine Phosphate 0.25 mg/kg
  Other Names: PQ
  Arms: 6Days Artemether/Lumefantrine+Primaquine
Other: Placebo — Aqueous solution prepared to mimic the taste of the intervention drug.
  Other Names: Placebo for Artemether Lumefantrine + Primaquine Phosphate
  Arms: 3 Days Artemether-Lumefantrine + Placebo

SUMMARY:
This clinical trial evaluates the advantage of prolonging the therapeutic life span of Artemether-lumefantrine from 3 days to 6 days, and addition of single low dose of Primaquine 0.25mg/kg. The study will have two arms, one that will receive standard treatment of uncomplicated malaria with Artemether-lumefantrine, and the other arm will receive the prolonged dose of 6 days together with single low dose primaquine. This approach is expected to provide strategies for malaria control in an era of imminent Plasmodium falciparum resistance.

DETAILED DESCRIPTION:
Despite documented high cure rates of ACT in Tanzania, and Africa elsewhere, clinical trials conducted in Tanzania with Swedish International Development cooperation Agency (SIDA) and Swedish Research Council support, provide evidence for in vivo selection of lumefantrine tolerant/resistant parasites among recurrent infections. Similarly, molecular epidemiology studies from Bagamoyo District, Tanzania, have shown temporal selection of lumefantrine associated genetic tolerance/resistance markers in the parasite population following wide scale use of Artemether-lumefantrine, but without signs of compromised treatment efficacy.

During the last decade, and despite the documented rapid microscopy determined parasite clearance of artemether-lumefantrine in Bagamoyo District, interest has developed in understanding the observation of high residual polymerase chain reaction (PCR) determined positivity rate on day 3 after supervised artemether-lumefantrine treatment in the magnitude of almost 30% in previous assessments from 2015. Using deep sequencing approaches studies have recently detected PCR determined delayed parasite clearance curves in P. falciparum sub-populations in Bagamoyo District. The clearance times by PCR of these sub-populations were similar to artemisinin resistant parasites in Myanmar as assessed by microscopy, but the former did, importantly, not harbor any of the described mutations in Kelch13 propeller associated with artemisinin resistance. However, these Tanzanian parasite sub-populations need to be further studied and characterized since they may provide important clues to the understanding of artemisinin survival strategies among the East African P. falciparum parasite population.

Taken together, longitudinal clinical and molecular data described above from Tanzania, East Africa, extending from pre-ACT implementation, (before 2006), to a decade of wide scale artemether-lumefantrine use in Bagamoyo district, provide evidence for declining susceptibility to ACT, both to artemether and lumefantrine, among the P. falciparum population. These parasites ("last man standing") that survived 10 years of ACT exposure have indeed shown excellent survival instincts and may thus be particularly resistant prone. However, if P. falciparum resistance to ACT develops in Africa, this will have devastating effects on malaria morbidity and mortality and may swiftly ruin the improvements the global malaria community achieved during the past decade with ACT as a key component for success.

Based on the above the investigators suggest prolonged treatment with ACT and addition of transmission blocking treatment using a single low dose of primaquine administered on the last day of ACT treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 1 year and less than 65 years.
2. Weight 10 kg and above;
3. Body temperature ≥37.5°C or history of fever in the last 24 hours;
4. Microscopy determined asexual P. falciparum mono-infection regardless of parasitemia
5. Normal - corrected QT Interval in Baseline ECG of less than 440ms in male and 460ms in females

Exclusion Criteria:

1. Symptoms/signs of severe malaria or danger signs;
2. Pregnancy, Breastfeeding or unwilling to practice birth control during participation in the study.
3. Known allergy to study medications;
4. Hb <8 g/dl;
5. Reported antimalarial intake within last 2 weeks;
6. On regular medication, which may interfere with antimalarial pharmacokinetics and
7. Blood transfusion within last 90 days.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2018-02-17 (Actual)

PRIMARY OUTCOMES:
Parasite Clearance Times | 5 Days
  Proportion of PCR detectable parasitemia on Day 5
Parasite Clearance Times | 7 Days
  Proportion of PCR detectable parasitemia on Day 7

SECONDARY OUTCOMES:
Gametocyte Clearance | 42 Days
  PCR determined gametocyte carriage/clearance times
Cure Rate | 28 Days
  Crude and PCR corrected cure rates by day 28
Genetic Markers of Drug Resistance | 6 Days
  Selection of genetic drug resistance markers during the early treatment phase
Pharmacokinetics | 7 Days
  Area under the plasma concentration versus time curve (AUC) of Artemether-lumefantrine
Peak Plasma Concentration (Cmax) | At hours, -1, 0 ,2 ,4 ,12, 24, 36, 40, 48, 52, 60, 72, 84, 88, 96, 100, 108,120, 132, 134, 136 ,144, 168, 192, 240, 336, 504 and 672
  Peak Plasma Concentration (Cmax) of Lumefantrine measured for 28 days
Day 7 plasma lumefantrine | 7 Days
  Day 7 plasma lumefantrine concentrations in the respective arms

OTHER OUTCOMES:
Fever Clearance Time | 7 Days
  This will assess the rate of clearance of fever after initiation of treatment
Incidence of Treatment-Emergent Adverse Events (Safety and tolerability) | Baseline and day 7
  Incidence of prolonged Corrected QT interval in ECG measures at day 7
Incidence of Severe anemia | baseline to day 7, 14, 28, 42
  Proportion of Severe anemia as measured by hemoglobin baseline to day 7, 14, 28, 42
Incidence of Biochemistry parameters derangements | Baseline and day 7
  Proportions of biochemistry parameters (ALAT, ASAT, Bilirubin and Creatinine) outside the normal range .

CONTACTS AND LOCATIONS:
Overall Officials: Lwidiko E Mhamilawa, MD, Principal Investigator — Muhimbili University of Health and Allied Sciences; Andreas Martensson, PhD, Study Chair — Uppsala University
Locations (2):
- Tanzania (2):
  - Fukayosi Dispensary, Bagamoyo, Coast Region
  - Yombo Dispensary, Bagamoyo, Yombo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sisowath C, Stromberg J, Martensson A, Msellem M, Obondo C, Bjorkman A, Gil JP. In vivo selection of Plasmodium falciparum pfmdr1 86N coding alleles by artemether-lumefantrine (Coartem). J Infect Dis. 2005 Mar 15;191(6):1014-7. doi: 10.1086/427997. Epub 2005 Feb 8. PMID 15717281
- [Background] Martensson A, Stromberg J, Sisowath C, Msellem MI, Gil JP, Montgomery SM, Olliaro P, Ali AS, Bjorkman A. Efficacy of artesunate plus amodiaquine versus that of artemether-lumefantrine for the treatment of uncomplicated childhood Plasmodium falciparum malaria in Zanzibar, Tanzania. Clin Infect Dis. 2005 Oct 15;41(8):1079-86. doi: 10.1086/444460. Epub 2005 Sep 13. PMID 16163624
- [Background] Malmberg M, Ngasala B, Ferreira PE, Larsson E, Jovel I, Hjalmarsson A, Petzold M, Premji Z, Gil JP, Bjorkman A, Martensson A. Temporal trends of molecular markers associated with artemether-lumefantrine tolerance/resistance in Bagamoyo district, Tanzania. Malar J. 2013 Mar 18;12:103. doi: 10.1186/1475-2875-12-103. PMID 23506218
- [Background] Mideo N, Bailey JA, Hathaway NJ, Ngasala B, Saunders DL, Lon C, Kharabora O, Jamnik A, Balasubramanian S, Bjorkman A, Martensson A, Meshnick SR, Read AF, Juliano JJ. A deep sequencing tool for partitioning clearance rates following antimalarial treatment in polyclonal infections. Evol Med Public Health. 2016 Jan 27;2016(1):21-36. doi: 10.1093/emph/eov036. PMID 26817485
- [Background] Mwaiswelo R, Ngasala BE, Jovel I, Gosling R, Premji Z, Poirot E, Mmbando BP, Bjorkman A, Martensson A. Safety of a single low-dose of primaquine in addition to standard artemether-lumefantrine regimen for treatment of acute uncomplicated Plasmodium falciparum malaria in Tanzania. Malar J. 2016 Jun 10;15:316. doi: 10.1186/s12936-016-1341-3. PMID 27287612
- [Background] R. Mwaiswelo, B. Ngasala, I. Jovel, W. Xu, and M. Malmberg, "Occurrence of day 3 submicroscopic Plasmodium falciparum parasitemia before and after implementation of artemether-lumefantrine treatment policy in Tanzania .," Dar Es Salaam, 2016
- [Background] Dondorp AM, Nosten F, Yi P, Das D, Phyo AP, Tarning J, Lwin KM, Ariey F, Hanpithakpong W, Lee SJ, Ringwald P, Silamut K, Imwong M, Chotivanich K, Lim P, Herdman T, An SS, Yeung S, Singhasivanon P, Day NP, Lindegardh N, Socheat D, White NJ. Artemisinin resistance in Plasmodium falciparum malaria. N Engl J Med. 2009 Jul 30;361(5):455-67. doi: 10.1056/NEJMoa0808859. PMID 19641202
- [Background] Ariey F, Witkowski B, Amaratunga C, Beghain J, Langlois AC, Khim N, Kim S, Duru V, Bouchier C, Ma L, Lim P, Leang R, Duong S, Sreng S, Suon S, Chuor CM, Bout DM, Menard S, Rogers WO, Genton B, Fandeur T, Miotto O, Ringwald P, Le Bras J, Berry A, Barale JC, Fairhurst RM, Benoit-Vical F, Mercereau-Puijalon O, Menard D. A molecular marker of artemisinin-resistant Plasmodium falciparum malaria. Nature. 2014 Jan 2;505(7481):50-5. doi: 10.1038/nature12876. Epub 2013 Dec 18. PMID 24352242
- [Background] Witkowski B, Amaratunga C, Khim N, Sreng S, Chim P, Kim S, Lim P, Mao S, Sopha C, Sam B, Anderson JM, Duong S, Chuor CM, Taylor WR, Suon S, Mercereau-Puijalon O, Fairhurst RM, Menard D. Novel phenotypic assays for the detection of artemisinin-resistant Plasmodium falciparum malaria in Cambodia: in-vitro and ex-vivo drug-response studies. Lancet Infect Dis. 2013 Dec;13(12):1043-9. doi: 10.1016/S1473-3099(13)70252-4. Epub 2013 Sep 11. PMID 24035558
- [Background] Straimer J, Gnadig NF, Witkowski B, Amaratunga C, Duru V, Ramadani AP, Dacheux M, Khim N, Zhang L, Lam S, Gregory PD, Urnov FD, Mercereau-Puijalon O, Benoit-Vical F, Fairhurst RM, Menard D, Fidock DA. Drug resistance. K13-propeller mutations confer artemisinin resistance in Plasmodium falciparum clinical isolates. Science. 2015 Jan 23;347(6220):428-31. doi: 10.1126/science.1260867. Epub 2014 Dec 11. PMID 25502314
- [Background] Malmberg M, Ferreira PE, Tarning J, Ursing J, Ngasala B, Bjorkman A, Martensson A, Gil JP. Plasmodium falciparum drug resistance phenotype as assessed by patient antimalarial drug levels and its association with pfmdr1 polymorphisms. J Infect Dis. 2013 Mar 1;207(5):842-7. doi: 10.1093/infdis/jis747. Epub 2012 Dec 5. PMID 23225895
- [Background] Linder E, Lundin M, Thors C, Lebbad M, Winiecka-Krusnell J, Helin H, Leiva B, Isola J, Lundin J. Web-based virtual microscopy for parasitology: a novel tool for education and quality assurance. PLoS Negl Trop Dis. 2008;2(10):e315. doi: 10.1371/journal.pntd.0000315. Epub 2008 Oct 22. PMID 18941514
- [Background] Lundin M, Szymas J, Linder E, Beck H, de Wilde P, van Krieken H, Garcia Rojo M, Moreno I, Ariza A, Tuzlali S, Dervisoglu S, Helin H, Lehto VP, Lundin J. A European network for virtual microscopy--design, implementation and evaluation of performance. Virchows Arch. 2009 Apr;454(4):421-9. doi: 10.1007/s00428-009-0749-3. Epub 2009 Mar 12. PMID 19280223
- [Background] Aydin-Schmidt B, Xu W, Gonzalez IJ, Polley SD, Bell D, Shakely D, Msellem MI, Bjorkman A, Martensson A. Loop mediated isothermal amplification (LAMP) accurately detects malaria DNA from filter paper blood samples of low density parasitaemias. PLoS One. 2014 Aug 8;9(8):e103905. doi: 10.1371/journal.pone.0103905. eCollection 2014. PMID 25105591
- [Background] Cook J, Aydin-Schmidt B, Gonzalez IJ, Bell D, Edlund E, Nassor MH, Msellem M, Ali A, Abass AK, Martensson A, Bjorkman A. Loop-mediated isothermal amplification (LAMP) for point-of-care detection of asymptomatic low-density malaria parasite carriers in Zanzibar. Malar J. 2015 Jan 28;14:43. doi: 10.1186/s12936-015-0573-y. PMID 25627037
- [Background] Aydin-Schmidt B, Morris U, Ding XC, Jovel I, Msellem MI, Bergman D, Islam A, Ali AS, Polley S, Gonzalez IJ, Martensson A, Bjorkman A. Field Evaluation of a High Throughput Loop Mediated Isothermal Amplification Test for the Detection of Asymptomatic Plasmodium Infections in Zanzibar. PLoS One. 2017 Jan 17;12(1):e0169037. doi: 10.1371/journal.pone.0169037. eCollection 2017. PMID 28095434
- [Background] Xu W, Morris U, Aydin-Schmidt B, Msellem MI, Shakely D, Petzold M, Bjorkman A, Martensson A. SYBR Green real-time PCR-RFLP assay targeting the plasmodium cytochrome B gene--a highly sensitive molecular tool for malaria parasite detection and species determination. PLoS One. 2015 Mar 16;10(3):e0120210. doi: 10.1371/journal.pone.0120210. eCollection 2015. PMID 25774805
- [Background] Mlambo G, Vasquez Y, LeBlanc R, Sullivan D, Kumar N. A filter paper method for the detection of Plasmodium falciparum gametocytes by reverse transcription polymerase chain reaction. Am J Trop Med Hyg. 2008 Jan;78(1):114-6. PMID 18187793
- [Background] Schneider P, Reece SE, van Schaijk BC, Bousema T, Lanke KH, Meaden CS, Gadalla A, Ranford-Cartwright LC, Babiker HA. Quantification of female and male Plasmodium falciparum gametocytes by reverse transcriptase quantitative PCR. Mol Biochem Parasitol. 2015 Jan-Feb;199(1-2):29-33. doi: 10.1016/j.molbiopara.2015.03.006. Epub 2015 Mar 28. PMID 25827756
- [Background] Froberg G, Jornhagen L, Morris U, Shakely D, Msellem MI, Gil JP, Bjorkman A, Martensson A. Decreased prevalence of Plasmodium falciparum resistance markers to amodiaquine despite its wide scale use as ACT partner drug in Zanzibar. Malar J. 2012 Sep 11;11:321. doi: 10.1186/1475-2875-11-321. PMID 22966778
- [Background] Veiga MI, Ferreira PE, Bjorkman A, Gil JP. Multiplex PCR-RFLP methods for pfcrt, pfmdr1 and pfdhfr mutations in Plasmodium falciparum. Mol Cell Probes. 2006 Apr;20(2):100-4. doi: 10.1016/j.mcp.2005.10.003. Epub 2006 Feb 7. PMID 16460912
- [Background] Price RN, Uhlemann AC, Brockman A, McGready R, Ashley E, Phaipun L, Patel R, Laing K, Looareesuwan S, White NJ, Nosten F, Krishna S. Mefloquine resistance in Plasmodium falciparum and increased pfmdr1 gene copy number. Lancet. 2004 Jul 31-Aug 6;364(9432):438-447. doi: 10.1016/S0140-6736(04)16767-6. PMID 15288742
- [Derived] Mhamilawa LE, Wikstrom S, Mmbando BP, Ngasala B, Martensson A. Electrocardiographic safety evaluation of extended artemether-lumefantrine treatment in patients with uncomplicated Plasmodium falciparum malaria in Bagamoyo District, Tanzania. Malar J. 2020 Jul 14;19(1):250. doi: 10.1186/s12936-020-03309-2. PMID 32664948
- [Derived] Mhamilawa LE, Ngasala B, Morris U, Kitabi EN, Barnes R, Soe AP, Mmbando BP, Bjorkman A, Martensson A. Parasite clearance, cure rate, post-treatment prophylaxis and safety of standard 3-day versus an extended 6-day treatment of artemether-lumefantrine and a single low-dose primaquine for uncomplicated Plasmodium falciparum malaria in Bagamoyo district, Tanzania: a randomized controlled trial. Malar J. 2020 Jun 23;19(1):216. doi: 10.1186/s12936-020-03287-5. PMID 32576258
- See also: "WHO World Malaria Report 2015," Geneva, Switzerland, 2015 — http://apps.who.int/iris/bitstream/10665/200018/1/9789241565158_eng.pdf
- See also: WHO guidelines for the treatment of malaria 2015, 3rd Edition. Geneva, Switzerland, 2015 — http://apps.who.int/iris/bitstream/10665/162441/1/9789241549127_eng.pdf
- See also: PRESIDENT'S MALARIA INITIATIVE Tanzania Malaria Operational Plan FY 2015 — https://www.pmi.gov/docs/default-source/default-document-library/malaria-operational-plans/fy-15/fy-2015-tanzania-malaria-operational-plan.pdf?sfvrsn=3

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT03241901/Prot_SAP_ICF_000.pdf